CLINICAL TRIAL: NCT06659913
Title: Project 3/7; Increased Physical Activity for Body and Mind
Acronym: Project 3/7
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 245639
Record Dates: First submitted 2023-03-13; First posted 2024-10-26 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Mental Health Impairment
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: RCT
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): The participants in the exercise group will be encouraged to follow the Norwegian Health authority's recommendation of being physically active for an average of 60 minutes a day, but they will also be offered a three-part intervention as a supplement to ordinary treatment. Supervised exercise will be offered once a week and they're encouraged to perform two additional exercise sessions per week.
  Interventions: Behavioral: Exercise training
- Control group (Active Comparator): The control group will receive treatment as usual
  Interventions: Behavioral: Exercise training

INTERVENTIONS:
Behavioral: Exercise training — Session 1: Consist of high intensity interval training performed on spinning bikes. An exercise physiologist will supervise the participants to perform a light 10 min warm-up, followed by 4 min working periods (intervals) interspersed by 3 min active breaks. The intensity should be 85-95% of estimated peak heart rate, corresponding to approximately 16 on the Borg scale (17). There will be a maximum of 10 participants in each group, depending on how many patients who are recruited for each of the two inclusion periods.I In addition, participants are encouraged to participate in the physical education at school and encouraged to perform exercise during the weekend, either with their family or friends.

SUMMARY:
The association between adequate amount of physical activity and good health is well established and for children and young people, and sufficient physical activity is an important factor for normal growth and development. Contrary, physical inactivity is associated with higher symptom pressure of mental disorders. Adolescents with mental disorders report to be less active compare the general population, with potentially increased risk of health and lifestyle diseases. This project aims to provide new knowledge on the degree of physical activity, motivation for physical activity and subjective perception of health in adolescents in need of mental health care. Further, this project aim to provide possible solution on how to increase physical activity in this patient group. Thus, this project has the potential to impact future guidelines for mental health services for adolescents in need of mental health care.

DETAILED DESCRIPTION:
Children and adolescents are recommended to perform at least 60 minutes per day of moderate-to-vigorous intensity. Further the guidelines state that children and adolescents should, incorporate vigorous-intensity aerobic activities that strengthens muscle and skeleton at least three times a week. High intensity training has been reported to have a positive effect on mental health variables in adults with mental disorders. However, the literature lacks studies on how this exercise regime affect the degree of and motivation for physical activity in inactive adolescents suffering from mental disorders. There are few studies, especially Norwegians, that have been done on this field, and more research on how we can follow up on these guidelines is urgently needed. This project is divided into three research questions:

1. Is it possible to increase the motivation for and degree of physical activity by a 3-joint training intervention including 1) Supervised exercise training group, 2) School based training supported by teacher in physical education, 3) Homebased training supported by caregivers, in adolescence between 12-17 years of age with low physical activity level referred to CAP clinic?
2. Compared to treatment as usual; is it possible to reduce the psychiatric symptom pressure and increase quality of life in adolescents at CAP clinic, by a 12-week training intervention including 1) Supervised exercise training group, 2) School based training supported by teacher in physical education, 3) Homebased training supported by caregivers?
3. Are physical activity level, psychiatric symptom pressure, and quality of life changed 6 months post exercise intervention (after 12-weeks) in adolescents at CAP clinic?

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria is low levels of physical activity, defined as not participating in any sport activity and/or drop-out of PE in school.

Exclusion Criteria:

Exclusion criteria are patients with a serious eating disorder or other health condition where exercise is not recommended.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Estimated)
Dates: Start 2023-04-13 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Physical activity level | after 12 weeks intervention
  Obejctively measured total physical activity level

SECONDARY OUTCOMES:
Psychiatric symptom pressure and quality of life | after 12 weeks intervention
  Psychiatric symptom pressure and quality of life will be measured using questionaires
Physical activity level, Psychiatric symptom pressure and quality of life | 6 months after intervention
  Same outcome as Outcome 1 and Outcome 2 post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Dorthe Stensvold Stensvold, Principal Investigator — Dorthe Stensvold, Professor, NTNU
Locations (1):
- Norwegian University of Science and Technology, Faculty of medicine, Department of circulation and medical imaging,, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: Undecided